CLINICAL TRIAL: NCT06762860
Title: The Effect of Intravenous Granisetron Versus Intravenous Dexmedetomidine on Shivering Following Spinal Anesthesia in the Cesarean Section. a Randomized Controlled Comparative Trial .
Brief Title: Intravenous Granisetron Vs Dexmedetomidine on Postspinal in the Cesarean Section.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Mennatallah Mamdouh, lecturer at faculty of medicine -Minia University , Menna.Mamdouh@mu.edu.eg, Minia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: postspinal shivering
Record Dates: First submitted 2024-12-03; First posted 2025-01-08 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-01

CONDITIONS: Postspinal Shivering
Keywords: shivering after spinal anesthesia in cesarean section
MeSH Terms: interventions — Dexmedetomidine; Granisetron

STUDY DESIGN:
Intervention Model Description: Group C: Patients in this group will receive 10 ml normal saline (0.9%) over 10minutes immediately after clamping of the cord (control group).
  Group D: Patients in this group will receive (0.3 ug/kg) intravenous Dexmedetomidine added to normal saline to get 10 ml of colorless solution and injected over 10 minutes after clamping of the cord.
  Group G: Patients in this group will receive 3 mg intravenous Granisetron added to normal saline to get 10 ml of colorless solution and injected over 10 minutes immediately after clamping of the cord.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Dexmedetomidine Group (Active Comparator): Patients in this group will receive (0.3 ug/kg) intravenous dexmedetomidine added to normal saline to get 10 ml of colorless solution and injected over 10 minutes after clamping of the cord.
  Interventions: Drug: Dexmedetomidine
- Granisetron Group (Active Comparator): Patients in this group will receive 3mg intravenous Granisetron added to normal saline to get 10 ml of colorless solution and injected over 10 minutes immediately after clamping of the cord.
  Interventions: Drug: Granisetron
- Control Group (Placebo Comparator): Patients in this group will receive 10 ml normal saline 0.9% over 10 minutes immediately after clamping of the cord (placebo control group).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexmedetomidine — label sticker
  Arms: Dexmedetomidine Group
Drug: Granisetron — label sticker
  Arms: Granisetron Group
Other: Placebo — label sticker
  Arms: Control Group

SUMMARY:
The Aim of this study is to investigate and compare the efficacy of intravenous Dexmedetomidine (0.3 ug/kg) versus intravenous Granisetron (3 mg) in the prevention of shivering in parturient undergoing cesarean section under spinal anesthesia.

DETAILED DESCRIPTION:
Study groups:

Randomization will be done according to computer guided table with sealed closed envelopes prepared by the supervisor, All study drugs will be prepared by the supervisor. Each group will be 25 patients.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for cesarean section under spinal anesthesia.
* age : (20-45) years old.
* American Society of Anesthesia (ASA) physical status I, II.

Exclusion Criteria:

* Patient refusal.
* Contraindication to spinal anesthesia.
* BMI > 35 kg/m².
* Impaired renal, hepatic and cardiac function.
* Thyroid disease.
* Body temperature >38 °C or < 36.5 °C.

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-01-30 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
The incidence and severity of post spinal shivering. | every 10 minutes intraoperatively and every 15 minutes postoperatively for 4 hours
  -The Shivering will be graded on a scale Tsai and Chu [Tsai et al .,2001] : Grade 0= No shivering. Grade 1=Piloerection or peripheral vasoconstriction but no visible shivering. Grade 2=Muscular activity in only one muscle group. Grade 3=Muscular activity in more than one muscle group but not generalized. Grade 4=Shivering involving the whole body.

SECONDARY OUTCOMES:
change in the basal axillary temperature. | preoperatively, immediately after spinal block and at 5 ,15 ,30 ,45 minutes and at the end of surgery, then every 15 minutes for 4 hour postoperatively
  Changes in basal axillary temperature (Celsius (°C) scale) of the patient after administration of tested drugs.
change in the basal mean arterial blood pressure | preoperatively, immediately after spinal block and at 5 ,15 ,30 ,45 minutes and at the end of surgery, then every 15 minutes for 4 hour postoperatively.
  Changes in the basal non-invasive mean arterial blood pressure( millimetres mercury (mmHg)) of the patient after administration of tested drugs.
Change in the basal heart rate | preoperatively, immediately after spinal block and at 5 ,15 ,30 ,45 minutes and at the end of surgery, then every 15 minutes for 4 hour postoperatively.
  Change in the heart rate of the patient after administration of tested drugs (beat per minute)

CONTACTS AND LOCATIONS:
Locations (1):
- Minya University Faculty of Medicine, Minya, Egypt

IPD SHARING:
Plan to Share IPD: No